CLINICAL TRIAL: NCT06555692
Title: After Mastectomy in Breast Cancer Patients, Prospective and Retrospective Study to Evaluate the Clinical Effectiveness and Safety of Supercritical Carbon Dioxide Processed Acellular Dermal Matrix(SC DERM® Recon) in Breast Reconstruction
Brief Title: Evaluation of the Clinical Effectiveness and Safety of Acellular Dermal Matrix(SC DERM® Recon) in Breast Reconstruction
Acronym: SCderm
Status: Recruiting | Type: Observational
Sponsor: DOF Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-01-002
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Female; Breast Reconstruction
Keywords: Acellular Dermal Matrix(ADM); Breast Reconstruction using implants and ADM

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: Among patients scheduled for total mastectomy due to the breast cancer, Female patients aged 20 to 69 who are willing to undergo immediate breast reconstruction using implants will be enrolled. The test group will be prospectively selected in 60 patients who undergo the breast reconstruction surgery applying with SC Derm(Inverstigational ADM processed by the supercritical technology).
  Interventions: Biological: Transplant acellular dermal matrix(ADM)
- Control Group: The control group will be retrospectively collected in 60 patients who underwent the breast reconstruction surgery applying with other ADM from the current medical records for one year of 2022.
  Among patients who underwent implant-based immediate breast reconstruction after total mastectomy, those who had the procedure between January 1, 2022, and December 31, 2022, and who completed at least 6 months of follow-up by June 2023 were included in the study.
  For this retrospective study, medical records of patients who met the inclusion and exclusion criteria were extracted. Data collection was carried out in the same manner as it would be for a prospective study.
  Interventions: Biological: Transplant acellular dermal matrix(ADM)

INTERVENTIONS:
Biological: Transplant acellular dermal matrix(ADM) — The principle of surgery is the pectoral muscle preservation (prepectoral) method and the subpectoral method (Breast Reconstruction using implants). After wrapping the implant with acellular dermal matrix(ADM), it is inserted into the breast and fixed to the underlying muscle or surrounding tissue depending on the situation.

SUMMARY:
This is the multi-centered, open, prospective and retrospective study of up to total 120 subjects in breast reconstruction surgery with applying acellular dermal matrix(ADM). The aim of the study is to ascertain any difference in the rate of complications between the test group of undergoing breast reconstruction with SC Derm and the control group of taking breast reconstruction with other ADM products.

DETAILED DESCRIPTION:
In South Korea, breast reconstruction surgery using implants or autologous abdominal tissue is commonly performed as the standard treatment to address the aesthetic and psychological needs of breast cancer patients who have undergone total mastectomies. In this procedure, acellular dermal matrix (ADM) is used to compensate for the skin deficit resulting from the removal of cancerous tissue. This clinical study is designed to ascertain whether there are differences in clinical efficacy, aesthetic outcomes, and safety in breast reconstruction surgery using ADM processed with supercritical carbon dioxide technology compared to other ADMs. The test group will be prospectively selected in 60 patients who undergo the breast reconstruction surgery applying with SC Derm(Inverstigational ADM processed by the supercritical technology). The control group will be retrospectively collected in 60 patients who underwent the breast reconstruction surgery applying with other ADM from the current medical records for one year of 2022.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 20 to 69 scheduled for total mastectomy
* Patients who are willing to undergo immediate breast reconstruction using implants.

Exclusion Criteria:

* Patients who have undergone organ transplantation and are currently taking immunosuppressive medication.
* Patients with mental conditions that could impact the conduct of the clinical study, such as alcohol or drug abuse.
* Patients who have participated in another clinical trial within 120 days prior to screening.
* Any other cases where the investigator deems the patient unsuitable for this clinical study.

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients who have undergone total mastectomy due to breast cancer from three primary university hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Breasts by Independent Investigator Using a 5-Point Likert Scale | 6 months after surgery
  Cosmetic outcome evaluation: Independent evaluation by two specialists for breast shape, size, symmetry, nipple position, and scar using standardized breast photos taken before surgery and at 6 months after surgery.
  Evaluation: Evaluate the score for each item using a 5 point Likert scale
  1. Shape : Very dissatisfied < Dissatisfied < Neutral < Satisfied < Very Satisfied
  2. Volume : Very dissatisfied < Dissatisfied < Neutral < Satisfied < Very Satisfied
  3. Symmetry : Very dissatisfied < Dissatisfied < Neutral < Satisfied < Very Satisfied
  4. Nipple-areolar Complex : Very dissatisfied < Dissatisfied < Neutral < Satisfied < Very Satisfied
  5. Scar : Very dissatisfied < Dissatisfied < Neutral < Satisfied < Very Satisfied

SECONDARY OUTCOMES:
Subject's Satisfaction Assessment | Beaseline to 6 months
  The patients' self-assessment of their satisfaction with the surgical outcomes at one month and 6 months visit of post-operation.
Baker's grade of capsular contracture | 6 months after surgery
  The occurrence of capsular contracture will be assessed clinically at the same follow-up visits (1 month and 6 months post-surgery).
  Grade I: Breast is normally soft and appears natural Grade II: Breast is a little firm but appears normal Grade III: Breast is firm and appears abnormal Grade IV: Breast is hard, painful, and appears abnormal
Complication Assessment | from the operation day to 6 months after surgery
  Evaluate the frequency and incidence rate of most commonly occurred complications of infection, skin necrosis, seroma, hematoma, implants removal.

CONTACTS AND LOCATIONS:
Overall Officials: Woojin Song, Ph.D, Principal Investigator — Soon Chun Hyang University
Locations (1):
- Soon Chun Hyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Polotto S, Bergamini ML, Pedrazzi G, et al. One-step prepectoral breast reconstruction with porcine dermal matrix-covered implant: a protective technique improving the outcome in post-mastectomy radiation therapy setting. Gland Surg 2020;9(2):219-228. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7225454/
- See also: Hagarty SE, et al. Decreased length of postoperative drain use, parental opioids, length of stay and complication rates in patients receiving meshed versus unmeshed ADM. Plast Reconstr Surg 2020; 145(4):889-897. — https://pubmed.ncbi.nlm.nih.gov/32221196/
- See also: Viezel-Mathieu A, Alnaif N, Aljerian A, et al.Acellualr dermal matrix-sparing direct-to-implant prepectoral breast reconstruction: A comparative study including cost analysis. Ann Plast Surg 2020;84(2):139-143. — https://pubmed.ncbi.nlm.nih.gov/31335468/
- See also: Nam SY, Youn D, Kim GH, et al. In vitro characterization of a novel human acellular dermal matrix (BellaCell HD) for breast reconstruction. Bioengineering (Basel) 2020;7(2):39. — https://pubmed.ncbi.nlm.nih.gov/32353944/
- See also: Heath, D.E. A Review of Decellularized Extracellular Matrix Biomaterials for Regenerative Engineering Applications. Regen. Eng. Transl. Med. 2019;5;155-166. — https://link.springer.com/article/10.1007/s40883-018-0080-0
- See also: Seo Y, Jung Y, Kim SH. Decellularized heart ECM hydrogel using supercritical carbon dioxide for improved angiogenesis. Acta Biomater. 2018; 67:270-281 — https://pubmed.ncbi.nlm.nih.gov/29223704/
- See also: Srivastava V, Basu S, Shukla VK. Seroma formation after breast cancer surgery: what we have learned in the last two decades. J Breast Cancer. 2012;15(4):373-380 — https://pubmed.ncbi.nlm.nih.gov/23346164/
- See also: Sforza M, Husein R, Atkinson C, Zaccheddu R. Unraveling Factors Influencing Early Seroma Formation in Breast Augmentation Surgery. Aesthet Surg J. 2017 Mar 1;37(3):301-307. — https://pubmed.ncbi.nlm.nih.gov/28207027/
- See also: A retrospective review of breast reconstruction outcomes comparing AlloDerm and DermaCELL. Heather Greig, Janine Roller, William Ziaziaris, Nancy Van Laeken. JPRAS Open, 2019 Jul;22:19-26 — https://pubmed.ncbi.nlm.nih.gov/32158893/